CLINICAL TRIAL: NCT00071032
Title: Functional Outcomes in Cardiovascular Patients Undergoing Surgical Hip Fracture Repair (FOCUS)
Brief Title: Safety and Effectiveness of Two Blood Transfusion Strategies in Surgical Patients With Cardiovascular Disease
Acronym: FOCUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey L Carson, MD, Jeffrey L Carson, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 159; U01HL073958-06 (NIH); U01HL073958 (NIH); U01HL074815 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Anemia; Hematologic Diseases; Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Thromboembolism; Pneumonia; Cerebrovascular Accident
Keywords: Blood Disease; blood transfusion
MeSH Terms: conditions — Anemia; Hematologic Diseases; Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Thromboembolism; Pneumonia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal (10 g/dL) Transfusion Strategy (Experimental): Transfusion strategy that maintains postoperative Hgb levels above 10 g/dL.
  Interventions: Biological: Liberal (10 g/dL) Transfusion Strategy
- 2 (Active Comparator): Symptomatic transfusion strategy, a more conservative strategy, in which blood transfusion is withheld until the patient develops symptoms of anemia.
  Interventions: Biological: Restrictive (Symptomatic) Transfusion Strategy

INTERVENTIONS:
Biological: Liberal (10 g/dL) Transfusion Strategy — This transfusion strategy will maintains postoperative Hgb levels above 10 g/dL. This threshold strategy will use enough red blood cell units to maintain Hgb levels at or above 10 g/dL through hospital discharge or up to 30 days after randomization.
  Arms: Liberal (10 g/dL) Transfusion Strategy
Biological: Restrictive (Symptomatic) Transfusion Strategy — Transfusion is withheld until the patient develops symptoms from anemia (i.e., chest pain or ECG changes thought to be ischemic, congestive heart failure, unexplained tachycardia or hypotension unresponsive to fluids) or until the hemoglobin level falls below 8 g/dL. Transfusion is permitted, but is not mandatory, if the hemoglobin level falls below 8 g/dL.
  Arms: 2

SUMMARY:
The purpose of this study is to compare liberal red blood cell transfusion therapy with restrictive red blood cell transfusion therapy in surgical patients with cardiovascular disease or risk factors.

DETAILED DESCRIPTION:
BACKGROUND:

Red blood cell transfusions are an extremely common medical intervention in both the United States and worldwide; over 14 million units of blood are transfused in the United States. Between 60 and 70 percent of all blood is transfused in the surgical setting. Despite the common use of red blood cell transfusions, the threshold for transfusion has not been adequately evaluated and is very controversial. A decade ago, the standard of care was to administer a peri-operative transfusion whenever the hemoglobin (Hgb) level fell below 10 g/dl (the "10/30 rule"). Concerns about the safety of blood, especially with respect to HIV and hepatitis, and the absence of data to support a 10 g/dl threshold led to the current standard of care, which is to administer blood transfusions based on the presence of symptoms, and not a specific Hgb/hematocrit level. However, there have not been any randomized clinical trials done with surgical patients that have tested the efficacy and safety of withholding blood until the patient develops symptoms, or the "10/30" approach to transfusion. Patients with underlying cardiovascular disease are at greatest risk of adverse effects from reduced Hgb levels.

DESIGN NARRATIVE:

This is a multi-center randomized trial to test the effectiveness of a transfusion strategy that maintains postoperative Hgb levels above 10 g/dl (liberal transfusion) in improving patient outcome. This will be compared to the restrictive (symptomatic) transfusion strategy in which blood transfusion is withheld until the patient develops symptoms of anemia or Hgb less than 8 g/dL. Participants will be randomly assigned to one of the two transfusion strategies. The liberal (10 g/dl) threshold strategy will use enough red blood cell units to maintain Hgb levels at or above 10 g/dl through hospital discharge. Restrictive (Symptomatic) transfusion strategy patients will receive red blood cell transfusions for symptoms of anemia, although transfusion is also permitted, but not required, if the Hgb level falls below 8 g/dl. Outcomes will include functional recovery (primary outcome: ability to walk 10 feet across a room without human assistance or death 60 days post-randomization), lower extremity activities of daily living and instrumental activities of daily living, survival up to 60-days and long-term, disposition (i.e., nursing home placement), and postoperative complications (e.g., myocardial infarction, unstable angina, or death in hospital, pneumonia, wound infection, thromboembolism, stroke).

Ambulation at 60 days is known to be highly predictive of ultimate functional outcome as well as of mortality at one year. Because inability to walk has such important implications for quality of life, and because it is a common problem, it far outweighs the small risk of viral infection or other complications from transfusion in elderly patients.

The trial will also evaluate the effect of transfusion threshold on postoperative risk of acute cardiac ischemia. The strategy will be to enhance surveillance for ischemic events by increasing the number of EKG and serum troponin measurements beyond those already called for in the original FOCUS protocol.

There is an ancillary study to the trial (R01 HL085706) to examine delirium as an outcome in a subsample of 139 patients. We will assess short-term (in hospital) and longer-term (after 30 days) severity of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone surgical repair for a hip fracture
* Has a postoperative Hgb level below 10 g/dL within three days of surgery
* Diagnosis of cardiovascular disease (e.g., coronary artery disease, congestive heart failure, stroke or transient ischemic attack, or peripheral vascular disease) or cardiovascular risk factors (e.g., diabetes mellitus, hypertension, hypercholesterolemia, tobacco use, or creatinine levels greater than 2.0 mg/dL)

Exclusion Criteria:

* Unable to walk prior to hip fracture
* Declines blood transfusions
* Suffered multiple traumas
* Pathologic fracture of the hip due to malignancy
* Clinically recognized acute myocardial infarction within the 30 days prior to study entry
* Previously participated in the trial and fractured the other hip
* Symptoms associated with anemia (e.g., ischemic chest pain) or actively bleeding at the time of randomization

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2016 (Actual)
Dates: Start 2003-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Carson, MD, Study Chair — University Medicine & Dentistry of NJ; Michael Terrin, Principal Investigator — University of Maryland, College Park
Locations (1):
- University Medicine & Dentistry of NJ, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Carson JL, Terrin ML, Magaziner J, Chaitman BR, Apple FS, Heck DA, Sanders D; FOCUS Investigators. Transfusion trigger trial for functional outcomes in cardiovascular patients undergoing surgical hip fracture repair (FOCUS). Transfusion. 2006 Dec;46(12):2192-206. doi: 10.1111/j.1537-2995.2006.01056.x. No abstract available. PMID 17176334
- [Result] Carson JL, Terrin ML, Noveck H, Sanders DW, Chaitman BR, Rhoads GG, Nemo G, Dragert K, Beaupre L, Hildebrand K, Macaulay W, Lewis C, Cook DR, Dobbin G, Zakriya KJ, Apple FS, Horney RA, Magaziner J; FOCUS Investigators. Liberal or restrictive transfusion in high-risk patients after hip surgery. N Engl J Med. 2011 Dec 29;365(26):2453-62. doi: 10.1056/NEJMoa1012452. Epub 2011 Dec 14. PMID 22168590
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Zhang J, Chen Z, He Y. Comparison of liberal versus restrictive transfusion strategies after hip surgery in patients with coronary artery disease: a post hoc analysis of the FOCUS trial. BMC Cardiovasc Disord. 2024 Sep 18;24(1):498. doi: 10.1186/s12872-024-04151-z. PMID 39294606
- [Derived] Meng L, Wang X, Carson JL, Schlussel Y, Shapses SA. Vitamin D Binding Protein and Postsurgical Outcomes and Tissue Injury Markers After Hip Fracture: A Prospective Study. J Clin Endocrinol Metab. 2023 Dec 21;109(1):e18-e24. doi: 10.1210/clinem/dgad502. PMID 37633261
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Carson JL, Sieber F, Cook DR, Hoover DR, Noveck H, Chaitman BR, Fleisher L, Beaupre L, Macaulay W, Rhoads GG, Paris B, Zagorin A, Sanders DW, Zakriya KJ, Magaziner J. Liberal versus restrictive blood transfusion strategy: 3-year survival and cause of death results from the FOCUS randomised controlled trial. Lancet. 2015 Mar 28;385(9974):1183-9. doi: 10.1016/S0140-6736(14)62286-8. Epub 2014 Dec 9. PMID 25499165

RESULTS

PARTICIPANT FLOW:
Groups:
- Liberal (10 g/dL) Transfusion Strategy: Transfusion strategy that maintains postoperative Hgb levels >= 10 g/dL
- Restrictive Strategy: Blood transfusion is withheld until the patient develops symptoms of anemia or at physician discretion of the hemoglobin level falls below 8 g/dL
Period: Overall Study
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Started | 1007 | 1009
Completed | 998 | 1001
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Missing Primary Outcome | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized subjects
Groups:
- Liberal (10 g/dL) Transfusion Strategy: Transfusion strategy that maintains postoperative Hgb levels above 10 g/dL.
  Liberal (10 g/dL) Transfusion Strategy: Maintains postoperative Hgb levels above 10 g/dL. This threshold strategy uses enough red blood cell units to maintain Hgb levels at or above 10 g/dL through hospital discharge or up to 30 days after randomization.
- Restrictive Strategy: Symptomatic transfusion strategy, a more conservative strategy, in which blood transfusion is withheld until the patient develops symptoms of anemia.
  Restrictive (Symptomatic) Transfusion Strategy: Transfusion is withheld until the patient develops symptoms from anemia (i.e., chest pain or ECG changes thought to be ischemic, congestive heart failure, unexplained tachycardia or hypotension unresponsive to fluids) or until the hemoglobin level falls below 8 g/dL. Transfusion is permitted, but is not mandatory, if the hemoglobin level falls below 8 g/dL.
- Total: Total of all reporting groups
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy | Total
Number analyzed (Participants) | 1007 | 1009 | 2016
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.8 (8.8) | 81.5 (9.0) | 81.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 757 | 770 | 1527
  Male | 250 | 239 | 489
Region of Enrollment [Number; unit: participants]
  United States | 609 | 613 | 1222
  Canada | 398 | 396 | 794
Cardiovascular Disease [Number; unit: participants] — History of coronary artery disease, congestive heart failure, cardiovascular disease, or peripheral vascular disease
  participants
    History of Cardiovascular Disease | 637 | 631 | 1268
    No History of Cardiovascular Disease | 370 | 378 | 748

OUTCOME MEASURES:

1. Primary Outcome: Inability to Walk 10 Feet or Across a Room Without Human Assistance or Death
Description: ascertained via telephone follow-up
Time Frame: 60 days after randomization
Measure: Number; unit: participants
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 998 | 1001
participants | 351 | 347
Statistical Analysis 1: Comparison: Liberal (10 g/dL) Transfusion Strategy vs Restrictive Strategy; Test type: Superiority or Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.84 to 1.22] — Liberal Arm (numerator) compared to Restrictive Arm (denominator)

2. Secondary Outcome: Myocardial Infarction, Unstable Angina, or Death for Any Reason
Time Frame: In-hospital
Measure: Number; unit: participants
Groups:
- Restrictive Strategy: Symptomatic transfusion strategy, in which blood transfusion is withheld until the patient develops symptoms of anemia or at physician discretion of the hemoglobin level falls below 8 g/dL
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 1005 | 1008
participants | 43 | 52
Statistical Analysis 1: Comparison: Liberal (10 g/dL) Transfusion Strategy vs Restrictive Strategy; Test type: Superiority or Other; Risk Difference (RD) = -0.9, 99% CI 2-sided [-3.3 to 1.6] — Liberal Arm (numerator) compared to Restrictive Arm (denominator)

3. Secondary Outcome: Mortality at 30 Days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 995 | 1000
Participants | 52 | 43

4. Secondary Outcome: Mortality at 60 Days
Time Frame: 60 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 998 | 1001
Participants | 76 | 66

5. Secondary Outcome: Composite Outcomes (a) Death, Myocardial Infarction, or Pneumonia and b) Death, Myocardial Infarction, Pneumonia, Thromboembolism, or Stroke
Time Frame: In-hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 1005 | 1007
Participants
  Death, myocardial infarction, or pneumonia | 89 | 90
  Death, MI, pnuemonia, thromboembolism or stroke | 103 | 94

6. Secondary Outcome: Myocardial Infarction
Time Frame: In-hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 1005 | 1008
Participants | 23 | 38

7. Secondary Outcome: Postoperative Complications (e.g., Wound Infection, Thromboembolism, Stroke)
Time Frame: In hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 1005 | 1007
Participants
  Wound Infection | 14 | 8
  Thromboembolism | 12 | 8
  Stroke | 8 | 3

8. Secondary Outcome: Disposition Status (i.e., Nursing Home Placement)
Description: Nursing Home Residence
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 996 | 1001
Participants | 137 | 161

9. Secondary Outcome: Function - Lower Extremity Activities of Daily Living,at 30 Days
Description: Using the Functional Status Index, score range 0 to 11, higher scores indicate greater dependency
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 472 | 507
score on a scale | 7.3 (4.0) | 7.4 (5.9)

10. Secondary Outcome: Function - Instrumental Activities of Daily Living, at 30 Days
Description: Using the Older Americans Resources and Services Functional Assessment Questionnaire, score range from 0 to 4, higher scores indicating greater dependency
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 437 | 450
score on a scale | 3.9 (0.5) | 3.9 (0.4)

11. Secondary Outcome: Function - Fatigue/Energy, at 30 Days
Description: Using the Functional Assessment of Chronic Illnesses Therapy-Fatigue, score range from 0 to 52, higher scores indicating greater level of energy
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 456 | 459
score on a scale | 38.7 (7.7) | 38.6 (7.6)

12. Secondary Outcome: Function - Lower Extremity Activities of Daily Living. at 60 Days
Description: Scale range 0 to 11, higher scores indicate greater dependency
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 523 | 553
score on a scale | 5.1 (4.2) | 5.1 (4.3)

13. Secondary Outcome: Function - Instrumental Activities of Daily Living, at 60 Days
Description: Scale range 0 to 11, higher scores indicate greater dependency
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 389 | 411
score on a scale | 3.7 (0.8) | 3.7 (0.9)

14. Secondary Outcome: Function - Fatigue/Energy, at 60 Days
Description: Scale ranging from 0 to 52, higher scores indicating greater level of energy
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 544 | 525
score on a scale | 41.8 (7.3) | 42.3 (7.4)

15. Secondary Outcome: Length of Stay in Hospital for United States Participants
Time Frame: Days from randomization to discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 608 | 612
days | 3.67 (3.38) | 3.97 (3.89)

16. Secondary Outcome: Length of Stay in Hospital for Canadian Participants
Time Frame: Days from randomization to discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Number analyzed (Participants) | 397 | 394
days | 12.03 (9.31) | 12.70 (9.48)

ADVERSE EVENTS:
Time Frame: Up to 60 days following randomization
Description: Medical events were captured during hospitalization (up to 30 days); mortality was determined at 60 days. There were a total of 2016 Number of Participants at Risk (1007 in the "Liberal Strategy" and 1009 in the "Restrictive Strategy" Arms/Groups), however, the number at risk was not the same for all events due to some missing data.
Groups:
- Liberal (10 g/dL) Transfusion Strategy: Transfusion strategy that maintains post randomization Hgb levels >= 10 g/dL
Arm/Group | Liberal (10 g/dL) Transfusion Strategy | Restrictive Strategy
Serious Adverse Events (participants affected / at risk) | 76/1007 | 66/1009
Other Adverse Events (participants affected / at risk) | 0/1007 | 0/1009
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Liberal (10 g/dL) Transfusion Strategy (N=1007) | Restrictive Strategy (N=1009)
Death at 60 days (General disorders) | 76/998 (76) | 66/1001 (66) — Detected via telephone follow-up
Myocardial Infarction (Cardiac disorders) | 23/1005 (23) | 38/1008 — during hospitalization (up to 30 days)
Unstable Angina (Cardiac disorders) | 2/1005 (2) | 3/1008 (3) — during hospitalization (up to 30 days)
Congestive Heart Failure (Cardiac disorders) | 27/1005 (27) | 35/1007 (35) — during hospitalization (up to 30 days)
Stroke (Vascular disorders) | 8/1005 (8) | 3/1007 (3) — during hospitalization (up to 30 days)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes